CLINICAL TRIAL: NCT04932772
Title: Abdominal Muscles Recovery Response to Kinesiotaping in Women With Postnatal Diastasis Recti: a Randomized Controlled Trial
Brief Title: Abdominal Muscles Recovery Response to Kinesiotaping in Women With Postnatal Diastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohammed Khalaf Sayed ElArabi, Demonstrator, Department of Physical Therapy for Women's health, Faculty of Physical Therapy, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003222
Record Dates: First submitted 2021-06-04; First posted 2021-06-21 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diastasis Recti

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (kinesiotaping group) (Experimental): include 24 women will receive kinesiotaping combined with abdominal exercise (2sessions /week for eight weeks).
  Interventions: Other: Kinesiotaping; Other: Abdominal Exercises
- Group B (abdominal exercise group) (Active Comparator): include 24 women will receive abdominal exercise only.
  Interventions: Other: Abdominal Exercises

INTERVENTIONS:
Other: Kinesiotaping — Technique: Include Rectus Abdominas Muscles (RAM), Oblique Abdominal Muscles (OAM). Tape will be applied on RAM using muscles technique from origin to insertion of muscle with a tension between15-35%. Band will be start on symphysis pubis with no tension and then women make stretch on the abdominal region by deep abdominal inspiration and will end at xyphoid process. Finally will perform on the right and left external oblique muscles the procedure will be start with no tension from bottom and of 6-12 ribs and then the hip will be place in flexion and rotation to opposite direction and the band will tape on pubic bone with tension between 15-35% (Kase et al., 2003).
  Other Names: KT Tape; Medical Tape
  Arms: Group A (kinesiotaping group)
Other: Abdominal Exercises — Women in group B will receive abdominal muscles exercise (2 sessions/ week) for eight weeks. This program will be applied in both group A and B. The women will repeat the same exercise program on other days as home routine. This program is proposed by Kamel and Yousif, 2017, as based on the literature (Kamel and Yousif, 2017), there is no golden standard exercise program for DRAM. Illustrations of the exercises will be provided, so that the women could repeat the same exercise program on other days as a home routine. All the exercises will be performed while the subject tied a scarf around her abdomen. The following proposed one included sit ups, reverse sit-ups, reverse trunk twists, and U-seat exercises (Fig. 5). Each exercise was repeated 20 times and was increased by four repetitions each week throughout the interventions. In addition, a respiratory rehabilitation maneuver to involve the abdominal muscles, especially the transverse abdominis will be performed.

SUMMARY:
This study aims to investigate abdominal muscle recovery in response to KT by using objective method for assessment as digital caliper, and waist circumference. KT technique will include rectus abdominis, internal and external oblique muscles among females after normal vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Age will range from 25-35 years.
2. All women give birth by normal vaginal delivery.
3. Diastasis recti more than 2.5 cm at any point along linea alba.
4. Body mass index (BMI) less than 30 kg/m2.
5. After the end of Puerperium period i.e. after eight weeks postnatal.

Exclusion Criteria:

1. Women with skin over sensitivity to tape.
2. Women with abdominal skin diseases.
3. Abdominal hernia.
4. Previous cesarean section.
5. Multiple pregnancies more than 3 times.
6. Other abdominal or back operation.
7. Pregnancy related complications such as polyhydramnios, fetal macrostomia, diabetes, and hypertension.
8. Spinal disorders.
9. Lower limbs deformities.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Change from Abdominal Caliper at 8 weeks | Baseline and after 8 Weeks
  A nylon digital caliper (ISS carbon digital caliper, 0-75 / 0.01 mm) will be used to measure the inter-recti distance. The subject is positioned in a crook lying position on a portable floor mat without a pillow under her head, knees flexed to 90 degrees and hands relaxed on her thigh. Before the measurement the investigator marks the reference points with a tape measure and a removable pen on the abdominal wall: at the superior border of the umbilicus; 5 cm and 10 cm above the umbilicus; 2.5 cm and 5 cm below the umbilicus. Then while the subject was exhaling, she is instructed to lift her head and shoulders up, slide her hands towards her knees, until the inferior angle of scapulae are just off the mat. She maintains the curl-up for three seconds while the measurement was taken. Meanwhile the instructor palpated the medial borders of the rectus abdominis muscle, put the caliper to the measurement point and measured the inter-rectum diastasis (IRD).

SECONDARY OUTCOMES:
Change from Waist circumference at 8 weeks | Baseline and after 8 Weeks of training
  It will be used for evaluating the recovery of the abdominal muscles by using tape measurement according to the standard set out by the world health organization when women in standing position at end of normal expiration without compression on skin.
Change from Abdominal strength and endurance test one minute sit-up test at 8 weeks | Baseline and after 8 Weeks of training
  For assessment abdominal muscles endurance women will be lie down on exercise mat with knees bent and hand placed across the chest or on ears. The women feet are held by one physiotherapist. The examiner will ask the participant to go and simultaneously start stop watch. On listening the command the women will be lifting her upper body and touch knees with elbows and perform the same as many times as possible for next one minute. This procedure includes three trails of sit-ups test each for one minute, the final score will be the best of three attempts for assessment abdominal muscles strength. A 70° wood support was placed at the back of the patient.
Change from The Oswestry Low Back Pain Disability Questionnaire at 8 weeks | Baseline and after 8 Weeks of training
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluator's use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. The questionnaire include 10 sections. results will be calculated from the sum of the scores in each of 10 sections. Each section includes ratings from ZERO (no problem) to FIVE (complete disability). Section 1, pain intensity, section 2, personal care (washing, dressing etc.), section 3, lifting, section 4, walking, section 5, sitting, section 6, standing, section 7, sleeping, section 8, sex life (if applicable), section 9, social life, section 10, travelling. The score is calculated as: 100 x (sum of the scores in each section / number of sections scored X5). Minimum = 0, maximum = 100. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia M Kamel, Professor, Study Chair — Cairo University
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trial and after deidentification
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after study publication
Access Criteria: email: mohamedkhalaf.pt@o6u.edu.eg